CLINICAL TRIAL: NCT02061657
Title: Phase 1 Study of Misoprostol in Reducing Intraoperative Bleeding in Myomectomy Operations
Brief Title: Impact of Misoprostol on Blood Loss In Myomectomy Operations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ahmed Elnaggar, DR, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AIN-1111-MM
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-07

CONDITIONS: Leiomyoma
MeSH Terms: conditions — Leiomyoma | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myomectomy, rectal Misoprostol (Experimental): 25 patients undergoing myomectomy operation will receive two tablets of misoprostol (400 mcg) rectally two hours before the operation.
  Interventions: Drug: Misoprostol
- Myomectomy, Placebo (Active Comparator): Include 25 patients undergoing myomectomy operation will not receive misoprostol before the operation.
  Interventions: Drug: Placebo( for misoprostol)

INTERVENTIONS:
Drug: Misoprostol — 25 patients undergoing myomectomy operation will receive two tablets of misoprostol (400 mcg) rectally two hours before the operation
  Other Names: Cytotec
  Arms: Myomectomy, rectal Misoprostol
Drug: Placebo( for misoprostol) — Include 25 patients undergoing myomectomy operation will not receive misoprostol before the operation.
  Arms: Myomectomy, Placebo

SUMMARY:
The aim of this research work is to assess the effect of using single preoperative dose of rectal misoprostol in abdominal myomectomy operations on blood loss, duration of the operation and possible operative complications

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled study that will be conducted in Ain Shams University Maternity Hospital.

A total of 50 women scheduled to undergo myomectomy for symptomatic uterine myoma will be included in this study after taking their consent for this clinical trial after full explanation of the trial.

The total of 50 included patients will be divided into two groups: Group A (Study group;): will Include 25 patients undergoing myomectomy operation will receive two tablets of misoprostol (400 mcg) rectally two hours before the operation.Group B (Control group): will Include 25 patients undergoing myomectomy operation will not receive misoprostol before the operation.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal patients aged between 35 to 50 years old.
* Five or less symptomatic uterine myomas .
* Maximum diameter of the largest myoma is 6 cm .
* All myomas are subserous or intramural.
* Uterine size less than 24 weeks pregnancy

Exclusion Criteria:

* History of previous surgery.
* Allergy to Misoprostol.
* Hypertension.
* Cardiac and Pulmonary diseases.
* Patients who have bleeding disorders.
* Anemia (Hb < 10g %).
* Chronic endocrine or metabolic diseases such as Diabetes.
* Obesity (body mass index > 30 kg/m2).
* Cases that will require intraoperative conversion of myomectomy to hysterectomy.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
intraoperative blood loss | time from peritoneum opening till its closure around (1 Hour)

CONTACTS AND LOCATIONS:
Overall Officials: Abd El Mgeed I. Abd El Mgeed, Professor, Study Chair — Ain Shams University; Mohamed S. Ali, Professor, Study Director — Ain Shams University; Mohamed A. Abdel-Hafeez, Lecturer, Principal Investigator — Ain Shams University; Mina A. Yacoup, Fellow, Principal Investigator — Ain Shams University; Ahmed M. Elnaggar, Lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Maternity Hospital, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Abdel-Hafeez M, Elnaggar A, Ali M, Ismail AM, Yacoub M. Rectal misoprostol for myomectomy: A randomised placebo-controlled study. Aust N Z J Obstet Gynaecol. 2015 Aug;55(4):363-8. doi: 10.1111/ajo.12359. Epub 2015 Jul 14. PMID 26174128